CLINICAL TRIAL: NCT05981053
Title: Biological Effects in Consumers of Resveratrol-enriched Wine
Status: Completed | Type: Observational
Sponsor: PINER Pastor Manfredi Winery (Industry)
Collaborators: University of Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: #26122021
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Aging; Healthy Aging; Sarcopenia; Obesity
Keywords: Food Science & Technology; Epigenetic age; Biological aging; Body composition; Muscle mass; Fat mass; Wine enriched; Resveratrol; Wine and health; Antiaging wine
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Resveratrol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemical-Clinical Studies
  1. Ferritin
  2. Complete blood count w/Platelet count
  3. Mean cell volume
  4. RDW - Red Distribution Width
  5. ultrasensitive PCR
  6. Glycemia
  7. Creatinine
  8. albumin
  9. Alkaline Phosphatase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Wine enriched with Resveratrol — Wine enriched with Resveratrol
  Other Names: https://vinospiner.com.ar/

SUMMARY:
The objective of this clinical trial is to compare the health conditions of the participating population before and after an intervention with Resveratrol enriched wine.

The main questions it aims to answer are:

1. • The consumption of wine enriched with resveratrol could slow down or reverse the biological age ?
2. • The consumption of wine enriched with resveratrol could improve body composition fat mass / muscle mass ? The participants will be evaluated at the beginning and at the end of the clinical trial and will adopt only one change in their habits, that is, change the usual wine they consume with their meals for a wine enriched with resveratrol, in a moderate measure, 250 cc for men and 125 cc/day for women. The design of the study will be that each volunteer is their own control, pre and post intervention.

DETAILED DESCRIPTION:
Study objectives The objective of the study is to determine the possible relationship between the consumption of pure Malbec wine 100% enriched with pure resveratrol (150 mg/L of wine) ingested during meals, with biomarkers (oxidative stress, DNA damage, antioxidant defenses and chronic systemic inflammation in blood and urine), generated in the body by the damage produced by the oxidative stress of metabolism, age and chronic pathologies.

Procedures to follow

1. First visit A doctor will take details of your medical history, perform a complete physical examination, and explain the reasons for the study. If you meet the criteria and are eligible to be included in the study, you will only be told not to take dietary supplements or antioxidants and you will be seen again in the office two weeks later. At that time, you will be asked to carry out a blood laboratory analysis. These will be the Baseline Controls.
2. Visits 30, 60, 90 days:

   Each period between consultations is 30 days, during which time the participant follows a free diet. At the end of each month, you will go for a medical consultation and be given the resveratrol-enriched wine. In the 4th consultation (90 days) the procedure of the first consultation will be repeated. That is, Consultation + Fasting blood extraction.

   Observations of eventual adverse events will be recorded; the information will be recorded in the CRF (Clinical Research Form).

   All the instruments used will be used only for you (disposable material), to avoid all types of contagion or infection.
3. Biochemical Analysis Determination of analysis to perform on the samples obtained from venous blood, initial and final at 90 days.

   samples. Venous blood will be obtained with heparin at both moments according to the protocol, with a 12-h fast. Start and end at 90 days.

   Determinations. Analysis of oxidative damage, analysis of enzymatic antioxidant defenses, inflammatory response in polymorphonuclear cells (PMN), red blood cells, plasma, and general biochemical analysis will be performed.

   Biochemical-Clinical Studies
   1. Ferritin
   2. Complete blood count w/Platelet count
   3. Mean cell volume
   4. RDW - Red Distribution Width
   5. Ultrasensitive PCR
   6. Glycemia
   7. Creatinine
   8. albumin
   9. Alkaline Phosphatase
4. Body composition analysis The determination of the InBody analysis will be carried out at the beginning and at the end of the study.

Statistical analysis: The statistical analysis was performed using the Student t-test for paired samples (Prism 7.0, GraphPad, San Diego, CA, USA). The Student t-test was selected to evaluate a single biomarker at a time in eight series of paired data (D0 vs. D90 for chronological and DNAm PhenoAge, muscle mass and fat mass) for each patient before and after the intervention. Results with p < 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1.1 Minimum 40 years 1.2 Maximum 80 years
2. Gender 2.1 Male 2.2 Female
3. Habits 3.1 Regular wine consumers

Exclusion criteria

1. Age 1.1 under 40 years 1.2 over 80 years
2. Modifications in treatments during the clinical trial 2.1 Pharmacological 2.2 Non-Pharmacological.
3. Pregnant women.
4. Women in planned pregnancy during the study period.
5. Women in the lactation period.
6. Patients who have been hospitalized for an infectious disease.
7. Patients suffering from autoimmune pathologies.
8. Patients who have cancer.
9. Patients with gastrointestinal pathologies.
10. Patients who have a history of liver disease.
11. Patients who have a history of kidney disease.
12. Patients who have hematological disease.
13. Patients who present disorders of the disease of psychiatric origin.
14. Patients who have epilepsy.
15. Patients with allergies to the active principles of: 15.1 Wine 15.2 Resveratrol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and with risk factors of cardiovascular diseases
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Epigenetic age | 3 months
  DNAm Phenoage
InBody muscle mass | 3 months
  Body composition
Body composition | 3 months
  InBody fat mass

CONTACTS AND LOCATIONS:
Locations (1):
- Raul Francisco Pastor, Buenos Aires, Buenos Aires City, Argentina

REFERENCES:
- [Background] Levine ME, Lu AT, Quach A, Chen BH, Assimes TL, Bandinelli S, Hou L, Baccarelli AA, Stewart JD, Li Y, Whitsel EA, Wilson JG, Reiner AP, Aviv A, Lohman K, Liu Y, Ferrucci L, Horvath S. An epigenetic biomarker of aging for lifespan and healthspan. Aging (Albany NY). 2018 Apr 18;10(4):573-591. doi: 10.18632/aging.101414. PMID 29676998
- [Background] Pastor RF, Restani P, Di Lorenzo C, Orgiu F, Teissedre PL, Stockley C, Ruf JC, Quini CI, Garcia Tejedor N, Gargantini R, Aruani C, Prieto S, Murgo M, Videla R, Penissi A, Iermoli RH. Resveratrol, human health and winemaking perspectives. Crit Rev Food Sci Nutr. 2019;59(8):1237-1255. doi: 10.1080/10408398.2017.1400517. Epub 2017 Dec 5. PMID 29206058
- [Background] Pastor RF, Repetto MG, Lairion F, Lazarowski A, Merelli A, Manfredi Carabetti Z, Pastor I, Pastor E, Iermoli LV, Bavasso CA, Iermoli RH. Supplementation with Resveratrol, Piperine and Alpha-Tocopherol Decreases Chronic Inflammation in a Cluster of Older Adults with Metabolic Syndrome. Nutrients. 2020 Oct 15;12(10):3149. doi: 10.3390/nu12103149. PMID 33076345
- [Background] Fitzgerald KN, Hodges R, Hanes D, Stack E, Cheishvili D, Szyf M, Henkel J, Twedt MW, Giannopoulou D, Herdell J, Logan S, Bradley R. Potential reversal of epigenetic age using a diet and lifestyle intervention: a pilot randomized clinical trial. Aging (Albany NY). 2021 Apr 12;13(7):9419-9432. doi: 10.18632/aging.202913. Epub 2021 Apr 12. PMID 33844651